CLINICAL TRIAL: NCT07374887
Title: Short Term and Long Term Impact of Snoezelen Intervention and Reminiscence Therapy on Emotionality and Anxiety and the Dynamics of Their Change in Older Adults in Slovak Elderly Care Facilities
Brief Title: Impact of Snoezelen Intervention and Reminiscence Therapy on Seniors' Emotionality and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matej Bel University (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Diana Ďuricová, Principal Investigator, Matej Bel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UGA-06-DS-2025; 09I03-03-V05-00009 (Other Grant/Funding Number: Early stage grants - Matej Bel University in Banská Bystrica)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Emotionality; Anxiety
Keywords: emotionality; anxiety; elderly care facilities; older adult; snoezelen; reminiscence therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Snoezelen intervention (Experimental): The Snoezelen intervention involved 20 participants in the pre-test and re-test, and 16 participants in the re-test.
  Interventions: Other: Snoezelen intervention
- Reminiscence therapy (Experimental): The reminiscence therapy involved 20 seniors in the pre-test and re-test, and 18 seniors in the re-test II.
  Interventions: Other: Reminiscence therapy
- Control group (No Intervention): The control group did not participate in any of the interventions.

INTERVENTIONS:
Other: Reminiscence therapy — Reminiscence therapy included 13 activities (Ďuricová, 2026b). Activities were also incorporated into the daily schedule over a period of four weeks, during weekdays. In the Hriňovčan care facility, one activity was conducted daily (lasting 60 minutes) in the common room during designated morning and afternoon hours. The selection and implementation of the activities were strictly determined and organised. The older adults participated in a group setting, with 20 members. The activities were led by two social workers who participated in training with the author of the programme.
  Arms: Reminiscence therapy
Other: Snoezelen intervention — Snoezelen intervention included 28 originally designed activities (Ďuricová, 2026a). The ideas were incorporated into the daily schedule of older adults over a period of four weeks, during weekdays. In Hriňovčan care facility, within the Snoezelen environment, two consecutive activities were carried out daily (with a total duration of 60 minutes), during the afternoon hours. The selection of activities depended on the interests of the older adults. Their application was neither strictly determined nor rigidly organised. Clients participated in the Snoezelen sessions in groups of 5-6 members. The activities were facilitated by trained staff - social worker and instructor of social rehabilitation.
  Arms: Snoezelen intervention

SUMMARY:
The aim of the study is to verify and compare the short-term and long-term effectiveness (retention) of Snoezelen intervention and reminiscence therapy and to analyze the dynamics of changes in the level of emotionality and anxiety of seniors in experimental groups and the control group.

The main question is:

There are significant differences in the level of emotionality (negative and positive emotional states) and anxiety between the two experimental groups of seniors and the control group of seniors during the measurements (pre-test measurement vs. retest measurement I; pre-test measurement vs. retest measurement II; retest measurement vs. retest measurement II)?

Researchers will compare seniors receiving Snoezelen intervention, those receiving Reminiscence Therapy, and a control group without intervention to see if the interventions lead to measurable improvements in emotionality and anxiety.

Participants will take part in Snoezelen sessions, take part in Reminiscence Therapy sessions, complete pretest, retest and retest II assessments measuring emotionality and anxiety.

DETAILED DESCRIPTION:
The study was registered retrospectively due to a limited awareness of the requirement to register behavioural interventions at the time of its initiation in 2022/2023. Initially conceived as a small-scale exploratory project, formal trial registration was not deemed necessary in the early planning stages.

As a doctoral student and early-career researcher, I was initially unaware that behavioural intervention studies also require formal registration. However, as the research progressed and its scope and significance became clearer, I recognised the importance of fulfilling this requirement. Upon learning of the relevant guidelines, I promptly took the necessary steps to complete the registration.

Although registration occurred at a later stage, the study was carried out in accordance with a pre-specified protocol, strictly adhering to methodological and ethical standards-approved, for instance, by the Ethics Committee of Matej Bel University. The hypotheses, study design, and analysis plan were defined prior to data collection, thereby ensuring the rigour, integrity, and transparency of the research process.

Funded by the EU NextGenerationEU through the Recovery and Resilience Plan for Slovakia under the project No. 09I03-03-V05-0000.

ELIGIBILITY:
Inclusion Criteria:

* long-term residence in the facility,
* age over 62,
* willingness to participate,
* ability to participate (no severe cognitive or physical impairments)

Inclusion Criteria for Snoezelen:

* mentioned above
* participants who have undergone Reminiscence therapy as part of previous research

Exclusion Criteria:

* significant physical problems,
* significant mental health problems,
* unwillingness to participate

Min Age: 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The Scale of Emotional Habituation of Subjective Well-Being - SEHP (Džuka & Dalbert, 2002) | from participant enrollment to data collection after 8 months
  The Scale of Emotional Habituation of Subjective Well-Being - SEHP (Džuka & Dalbert, 2002) was used to examine the short-term effectiveness of the intervention programme. The self-esteem scale maps the frequency of experiencing positive and negative emotions, totalling 10. Negative emotional experiencing consists of six emotions such as anger, guilt, fear, pain, sadness, and shame, positive emotional experiencing consists of pleasure, physical freshness, joy, and happiness. The participants responded on a six-point scale (6 - almost always; 1 - almost never). The total score of negative emotions is the sum of negative emotions, and the total score of positive emotions is the sum of positive emotions (Džuka et al., 2021).
The Anxiety and Trait Anxiety Inventory - STAI (Spielberger et al., 1970, ed. Ruisel et al., 1980) | from participant enrollment to data collection after 8 months
  The Anxiety and Trait Anxiety Inventory - STAI (Spielberger et al., 1970, ed. Ruisel et al., 1980), specifically only the anxiety portion of the questionnaire, i.e., the Scale for the Measurement of Anxiety as a Condition, STAI X-1. This is the self-assessment portion of the questionnaire, which maps the degree of current experience of feelings of tension, tenseness, nervousness, fear, and apprehension. It contains 20 statements, some of which relate to the existence of these feelings and some of which relate to their absence. Seniors rated their experiencing on a four-point scale (4 - very, 1 - not at all). We based the norms on those presented in the manual by Ruisel et al. (1980).The result is a total score, which is obtained by summing the values on the scale taking into account reverse scaling. The range of the total score is 20-80.

SECONDARY OUTCOMES:
Reflection Questionnaire (Ďuricová, 2023) | one month
  This is a questionnaire that maps client satisfaction with activities. It includes three statements, with clients expressing their level of agreement on a three-point scale (agree - have no strong opinion - disagree) in the areas of: re participation, usefulness and disinterest in the activities. It also includes three incomplete sentences that seniors complete at will. Responses reflect what clients learned/how the activities helped them, what they liked most about the activities, what they would remove from the activities.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ďuricová, PhDr., Principal Investigator — Matej Bel University; Lenka Ďuricová, doc., Mgr., PhD., Study Director — Matej Bel University
Locations (1):
- Hriňovčan care facility for older adults, Hriňová, Slovakia 96205, Hriňová, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website of the organization where the research was conducted — https://www.zsshrinovcan.sk/